CLINICAL TRIAL: NCT06055582
Title: A Randomized Controlled Study to Compare Effects of Mango Ingestion on Glycemia (Glycemic Response, Continuous Glucose Monitoring and Fructosamine) Insulin Resistance and Body Composition in Patients With T2DM and Non-diabetic Subjects.
Brief Title: To Study the Effects of Mango Ingestion in T2DM and Non-diabetic Subjects.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diabetes Foundation, India (Other)
Collaborators: Indian Council of Medical Research (Other Government)
Responsible Party: Principal Investigator, Dr Anoop Misra, Director, Diabetes Foundation, India
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 5/9/1309/2020-Nut
Record Dates: First submitted 2023-07-19; First posted 2023-09-26 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Normoglycemia; T2DM (Type 2 Diabetes Mellitus)
Keywords: Insulin resistance; body composition; glycemic index
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Bread; Mangifera indica extract

STUDY DESIGN:
Intervention Model Description: Patients with T2DM and non-diabetic subjects were randomized into two food groups- mango and bread for 3 days, then after a 7 days washout period, the cross-over took place.
Masking Description: Patients were recruited from Fortis C-DOC OPD.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment - Mango (Other): Subjects in mango group will be further randomized into three different groups. Each group will be tested on a different variety of mango.
  Interventions: Dietary Supplement: Mango
- Controlled- Bread (Other): Subjects in bread group were given 81g (3 slices) harvest gold white bread as standard food in raw form.
  Interventions: Dietary Supplement: Bread

INTERVENTIONS:
Dietary Supplement: Bread — 81g (3 slices) harvest gold white bread as standard food.
  Arms: Controlled- Bread
Dietary Supplement: Mango — 250g of mango pulp of each mango variety was given to the subjects.
  Other Names: Safeda, Dushehri, Langra
  Arms: Treatment - Mango

SUMMARY:
T2DM patient will be recruited from endocrine OPD

1. Clinical History and Examination:

   1. General Physical Examination:

      * Height (cm)
      * weight (kg)
      * BMI (kg/m2)
      * Blood Pressure (mmHg)
   2. Anthropometry: Circumferences and skinfold thickness will be recorded for the patients in the following manner.

      Circumferences:
      * Waist circumference (cm)
      * Hip circumference (cm)
      * Mid-arm circumference (cm)
      * Mid-thigh circumference (cm)
   3. Skin fold thickness: Skin fold thickness will be measured by using (LANGE skin fold calipers) (to nearest of 1 mm) at the following sites

      * Biceps (mm)
      * Triceps (mm)
      * Thigh (mm)
      * Calf (mm)
      * Sub scapular (mm)
      * Supra-iliac (mm)
      * Anterior axillary fold. (mm)
2. Biochemical Test: The biochemical analysis will be done using ELISA kit or commercially available kits

   * Blood glucose (mg/dL)
   * HbA1c (%)
   * Serum insulin (μIU/mL)
   * Total Cholestrol (mg/dl)
   * Triglyceride (mg/dl)
   * Fructosamine (umol/L)
   * Adiponectin (µg/ml) -- HOMA-IR
3. Body Composition Analysis (TANITA)

DETAILED DESCRIPTION:
1. Phase I: Exploratory Acute Phase- Stratified randomized study

   * Study population: 2 groups; patients with T2DM and non-diabetic subjects n=45 (20 T2DM subject, 25 non-diabetic subjects).
   * Study groups: 3 groups; OGTT (n=5), mango (n=30), bread (n=10) Subjects in mango group will be further randomized into three different groups. Each group will be tested on a different variety of mango.

   Procedure for Phase I:

   After measuring baseline glucose level on empty stomach, three groups will be given their respective standardized food item and blood samples will be drawn every half an hour upto 2 hours of ingestion at (minutes): 0, 30, 60, 90 and 120. Fingertip capillary blood will be used for the estimation of blood glucose using a glucometer of contour brand.
2. Phase II: Exploratory Sub-Acute Phase- Two randomized cross over study

   * Study population: 2 groups; patients with T2DM and non-diabetic subjects, n=50 (25 in each study population group)
   * Study groups: 2 groups; mango (n=30), bread (n=20) Subjects in mango group will be further randomized into three different groups. Each group will be tested on a different variety of mango.

   Procedure for Phase II:
   1. Continuous glucose monitoring system (CGMS): It will be affixed for 3 days.
   2. The research team will be contacting the study subjects every day for any discomfort due to CGMS device or diet.
   3. On day 4 study subjects will be called to the study site and CGMS will be removed and data will be transferred to the study records.
   4. Study subjects will be asked to maintain a food diary and record the foods consumed during the entire period of 3 days.
   5. The subjects will also be asked to fill questionnaire of dietary assessment on Day 1 and Day 4 for per schedule of assessments.
3. Phase III: Confirmatory Chronic Phase- Randomized controlled parallel arm study

   * Study population: patients with T2DM, n=35
   * Study groups: 2 groups; mango (n=20), bread (n=15) Subjects in mango group will be further randomized into two different groups. Each group will be tested on a different variety of mango.

Procedure for Phase III:

Subjects will be given glucometers and will be asked to monitor blood glucose at fasting state and after standard breakfast meal at baseline, at day 30 and day 60 in both the study groups. The intermediate term effect of mango consumption and bread consumption will be assessed at baseline and at day 60 in terms of following investigations:

1. Dietary assessment
2. Physical activity (PA) assessment (GPAQ)
3. Blood pressure
4. Anthropometry measures
5. Body composition
6. Biochemical investigations

ELIGIBILITY:
Inclusion Criteria:

-For patients with diabetes: Stable glycemic control on metformin or sulfonylurea for past 3 months and without any major complications and HbA1C less than 8%

Exclusion Criteria:

* Acute infections and advanced end-organ damage
* History of hepatitis or pancreatitis, abnormal liver and renal functions
* Recent (<3 months) changes in weight
* Any known allergy to mangoes and bread
* Subjects with hypothyroidism
* On any drug causing weight gain or weight loss.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2022-02-11 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Outcome for all the phases will be as follows | Baseline, after six months of intervention
  Fasting glucose (mg/dL)
Postprandial blood glucose (mg/dL) | Baseline, after six months of intervention
Glycemic indices as per Continuous glucose monitoring system (CGMS) & HbA1c (%) | Baseline, after six months of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Anoop Misra, MD, Principal Investigator — Fortis CDOC Hospital
Locations (1):
- Fortis CDOC Hospital, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No